CLINICAL TRIAL: NCT02062697
Title: Pilot Study of the Lavage of the Uterine Cavity for the Diagnosis of Ovarian and Tubal Carcinoma and Their Premalignant Changes - LUDOC Study
Brief Title: Lavage of the Uterine Cavity for the Diagnosis of Ovarian and Tubal Carcinoma and Their Premalignant Changes.
Acronym: LUDOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Paul Speiser, Prof.MD,, Univ.Prof.MD., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK 1148/2011
Record Dates: First submitted 2014-01-20; First posted 2014-02-14 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Epithelial Cancer
Keywords: Neoplasms; Glandular and Epithelial; Ovarian Neoplasms; Ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ovarian Epithelial Cancer (Other): * Lavage of the Cavum uteri and proximal fallopian tubes
  * Liquid-PAP (Papanicolaou) smear
  Interventions: Procedure: Lavage of the Cavum uteri and proximal fallopian tubes; Procedure: Liquid-PAP smear

INTERVENTIONS:
Procedure: Lavage of the Cavum uteri and proximal fallopian tubes
  Other Names: MF 13005 (MADICOPLAST Catheter)
Procedure: Liquid-PAP smear

SUMMARY:
Epithelial Ovarian cancer (EOC) is the leading cause of death among gynaecologic malignancies in western civilized countries, with an estimated prevalence in Europe and the US of 752,600 in 2007 and 59,828 deaths annually.

State-of-the-art diagnostic tests for EOC include transvaginal ultrasonography and serum cancer antigen (CA-125) measurements; the specificity of these diagnostic tools however is low, and both tests are not effective enough at detecting EOC early enough to improve clinical outcomes. Definitive diagnosis of EOC still relies on histological or cytological confirmation. These findings underline the importance for an effective test for early detection of EOC.

In the current project we will obtain a lavage of the uterine cavity. It will be investigated whether cells from EOCs or genetic material from those cells can be detected in the lavage fluid.

Aim of this study:

There is a clear clinical need for a diagnosis test to detect EOC at an earlier stage.

DETAILED DESCRIPTION:
Epithelial Ovarian cancer is the leading cause of death among gynaecologic malignancies in western civilized countries, with an estimated prevalence in Europe and the US of 752,600 in 2007 and 59,828 deaths annually. Treatment and survival of the patients depend primarily on the stage of the disease. Of all EOC patients only 25% are diagnosed at an early stage while the tumour is confined to the pelvis. In these cases the five-year survival rate is 80% to 90% and the disease can often be cured by the combination of surgery and chemotherapy. Unfortunately, almost 75% of women affected have advanced stage disease with metastatic spread throughout the abdominal cavity or to retroperitoneal lymph nodes at the time of diagnosis; five-year survival rates drop to 10%-30% for advanced disease, despite maximum surgical effort and combination chemotherapy.

State-of-the-art diagnostic tests for EOC include transvaginal ultrasonography and serum cancer antigen (CA-125) measurements; the specificity of these diagnostic tools however is low, and both tests are not effective enough at detecting EOC early enough to improve clinical outcomes. Definitive diagnosis of EOC still relies on histological or cytological confirmation. These findings underline the importance for an effective test for early detection of EOC.

In the current project we will obtain a lavage of the uterine cavity. It will be investigated whether cells from EOCs or genetic material from those cells can be detected in the lavage fluid.

Aim of this study:

There is a clear clinical need for a diagnosis test to detect EOC at an earlier stage.

ELIGIBILITY:
Inclusion Criteria:

* suspected ovarian cancer
* verified ovarian cancer

Exclusion Criteria:

* pregnant
* incapacitated persons

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Detection of EOCs by mutation analysis in the lavage of the uterine cavity. | Day 1
  If the adnexal tumor removed turns out to be an EOC, mutation analysis will be carried out applying the sensitive massively parallel sequencing method published by Kinde et al. Mutations in the following genes will be analysed: AKT1, APC, ARID1A, BRAF, CTNNB1, CSMD3, CDKN2A, EGFR, FBXW7, FAT3, FGFR2, KRAS, MLL2, NRAS, PTEN, PIK3CA, PIK3R1, PPP2R1A, PIK3R, RNF43, and TP53.

SECONDARY OUTCOMES:
Detection of EOCs by mutation analysis of the liquid-based Pap smear. | Day 1
  Obtaining material from the uterine cervix by applying a liquid-based Pap smear technique to directly compare the two sampling techniques - Lavage and liquid-based Pap.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Speiser, Univ.Prof.Dr., Principal Investigator — Medical University Vienna, Dptm. of Obstetrics & Gynaecology
Locations (6):
- Medical University Vienna, Dptm. of Obstetrics & Gynaecology, Vienna, Austria
- University Hospitals Leuven - Department of Obstetrics and Gynaecology, Leuven, Belgium
- Charles University, Pilsen - Medical Faculty Hospital, Department of Obstetrics and Gynecology, Pilsen, Plzeň Region, Czechia
- Germany (3):
  - Charité University - Campus Virchow Clinic, Berlin
  - Klinik Essen Mitte (KEM), Essen
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg